CLINICAL TRIAL: NCT00985335
Title: Effectiveness of TheraNeem Lip Therapy of Common Symptoms of Herpes Simplex Labialis A Prospective Experimental Case Series (n=5)
Brief Title: Effectiveness of TheraNeem Lip Therapy for Herpes Simplex Labialis
Acronym: Neem
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sivarama Vinjamury, Professor, Southern California University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCU-09-VINJ004
Record Dates: First submitted 2009-08-28; First posted 2009-09-28 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Herpes Simplex
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External Application of Neem-based Cream (Experimental): Non Controlled, non-randomized, single group pilot study.
  Interventions: Other: Neem Based External Application Cream

INTERVENTIONS:
Other: Neem Based External Application Cream — Apply externally 3-4 times per day

SUMMARY:
This study intends to test the efficacy of the TheraNeem Lip Therapy balm for Herpes Simplex. The study will include a total of 5 people.

DETAILED DESCRIPTION:
Qualified candidates will be officially enrolled into the study within 24 hours of their subsequent outbreak of Herpes Simplex Labialis. They will be given all of the Neem Therapy products to use, and photographs and questionnaires will be taken to assess their progress.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has signs and symptoms of HSV-1 infection of less than 24 hours duration to the Southern California University of Health Sciences investigators
2. Participants ages 18-70 years
3. Confirmation of oral-circumoral herpes lesion will be made by a clinician in the presence of oral-circumoral lesion assumed to be HSV-1 for purposes of study
4. Subjects expressed willingness to comply with protocol
5. Subject will be willing to have the presenting lesion photographed twice
6. Subject sign a written informed consent, HIPPA disclosure, Experimental bill of rights

Exclusion Criteria:

1. History of past or present immunosuppressive condition, or currently taking immunosuppressive medication
2. History of adverse effects or allergies to any Neem based product or containing any of the other ingredients TheraNeem Lip Therapy: Organic Coconut Oil, Organic Beeswax, Organic Jojoba Oil, Shea Butter, Sesame Oil, Organic Neem Oil, , Essential Oil of Peppermint, Vitamin E (Tocopherol)
3. Signs of disseminated HSV illness
4. History of use of oral or topical antiviral agents within 10 days of screening and/or at start of study visit
5. Pregnancy or lactation
6. Psychiatric disorder
7. Inability to understand or follow the instructions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cold Sore Symptom Scale | Baseline and End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melany Meier, DC, Principal Investigator — Southern California University of Health Sciences; Sivarama Vinjamury, L.Ac, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- Southern California University of Health Science, Whittier, California, United States